CLINICAL TRIAL: NCT00440427
Title: A Randomized, Open-Label, Single-Dose Parallel Group Study of the Pharmacokinetic Profile, Safety, and Tolerability of 25- and 50-mg Desvenlafaxine Sustained Release (DVS SR) in Healthy Subjects
Brief Title: Study Evalutating the Pharmacokinetics (PK) and Safety of a Single Dose of Desvenlafaxine Sustained Release (DVS SR)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3151A2-1201
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: Desvenlafaxine Sustained Release (DVS SR)

SUMMARY:
To assess the initial pharmacokinetic profile of single doses of 25mg and 50 mg of DVS SR to healthy subjects.

ELIGIBILITY:
* Men or non-pregnant, non-lactating women
* Body mass index 18 - 30 kg/m2
* Body weight greater than or equal to 60kg

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2007-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Boston, Massachusetts, United States